CLINICAL TRIAL: NCT00677131
Title: Study of the Evaluation of Patient Education Efficacy: Reconstitution, Storage, and Administration of Oral Antibiotic Suspension From Powder Dosage Form at Pharmacy of National Taiwan University Hospital
Brief Title: Study of the Evaluation of Patient Education Efficacy in Pharmacy of National Taiwan University Hospital
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Li-Jiuan Shen, National Taiwan University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 200803049R
Record Dates: First submitted 2008-05-08; First posted 2008-05-13 (Estimated); Last update posted 2009-12-04 (Estimated); Status verified 2009-11

CONDITIONS: Infection
Keywords: pediatrics; antibiotics; patient education
MeSH Terms: conditions — Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Active Comparator): To read the package insert of the drug
  Interventions: Other: Reading the package insert of the drug
- 2 (Active Comparator): To read the education information provided by the Pharmacy of NTUH
  Interventions: Other: Reading the education information provided by the Pharmacy of NTUH
- 3 (Active Comparator): Oral education provided by the pharmacist
  Interventions: Other: Oral education provided by the pharmacist

INTERVENTIONS:
Other: Reading the package insert of the drug — package insert of the drug
  Arms: 1
Other: Reading the education information provided by the Pharmacy of NTUH — education information
  Arms: 2
Other: Oral education provided by the pharmacist — Oral education provided by the pharmacist
  Arms: 3

SUMMARY:
The primary purpose of this study is to evaluate the patient education efficacy of the pharmacists in National Taiwan University Hospital. We randomize patient family into one of the following three groups:

1. To read the package insert of the drug
2. To read the education information provided by Pharmacy of NTUH
3. Oral education provided by the pharmacist

Then we will evaluate the difference on patient knowledge of reconstitution, storage, and administration of oral antibiotic suspension from powder dosage form between these three groups.

DETAILED DESCRIPTION:
The primary purpose of this study is to evaluate the patient education efficacy of the pharmacists in National Taiwan University Hospital. We designed twelve questions about reconstitution, storage, and administration of oral antibiotic suspension from powder dosage form in a questionnaire. We will recruit pediatric patients who are prescribed one of the two oral antibiotics powder for suspension, Augmentin and Zithromax. We will randomize the family of these patients into one of the following three groups:

1. To read the package insert of the drug
2. To read the education information provided by Pharmacy of NTUH
3. Oral education provided by the pharmacist

Then we will ask them the twelve questions in the questionnaire and record their answer. Eventually, we will be able to compare the number of the correct answer, and to evaluate the difference on patient knowledge of reconstitution, storage, and administration of oral antibiotic suspension from powder dosage form between these three groups.

ELIGIBILITY:
Inclusion Criteria:

* Family of pediatric patient who is prescribed one of the two oral antibiotics granule for suspension, Augmentin and Zithromax, in NTUH

Exclusion Criteria:

* Family of pediatric patient who can not read Chinese

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2008-04; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Number of correct answer of questions that patient family make | At the end of education

SECONDARY OUTCOMES:
The type of the correct answer of question that patient family make | At the end of education

CONTACTS AND LOCATIONS:
Overall Officials: Li J Shen, doctor, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan